CLINICAL TRIAL: NCT00476424
Title: A Pharmacokinetic Study of Once Daily Efavirenz 400 mg Versus 600 mg in Thai HIV-1 Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Ministry of Education, Thailand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 081
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: once daily Efavirenz 400 mg; PK once daily Efavirenz 400 mg versus 600 mg; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 400 mg EFV
  Interventions: Drug: efavirenz
- 2 (Active Comparator): 600 mg EFV
  Interventions: Drug: efavirenz

INTERVENTIONS:
Drug: efavirenz — EFV 400 mg OD for 14 days EFV 600 mg OD for 14 days

SUMMARY:
A Pharmacokinetic study of once daily Efavirenz 400 mg versus 600 mg in Thai HIV-1 infected subjects.

DETAILED DESCRIPTION:
Efavirenz Pharmacokinetic evaluation supports once-daily dosing (T1/2 is 10-52 hours). The recommended dosage of efavirenz in combination with nucleoside reverse transcriptase inhibitor (NRTI) and/or protease inhibitor (PI) is 600mg orally, once daily.

In Thai populations, many ARV levels are very high. We believe that 600 mg efavirenz is too high for Thai people and would like to see the pharmacokinetic data and safety and efficacy of efavirenz at 400 mg.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age or older with HIV-1 infection
* Who are on stable PI-based highly active antiretroviral therapy and have HIV-1 RNA <50 copies/ml within 6 months.
* No active opportunistic infection.
* Sexually active subjects must be willing to use an effective form of birth control.
* Able to provide written informed consent.

Exclusion Criteria:

* Pregnant or breast-feeding females are excluded.
* Inability to understand the nature and extent of the study and the procedures required.
* ALT/ AST more than 5x upper limit
* Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of concomitant medication that may interfere with the pharmacokinetics of efavienz
* History of sensitivity/idiosyncrasy to the drug or chemically related compounds which may be employed in the study.
* Active drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Assess whether the low dose efavirenz is not inferior to the standard dose of efavirenz in terms of plasma concentration | 6 weeks

SECONDARY OUTCOMES:
Access efavirenz plasma level after discontinuation of this medication | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)
Locations (1):
- The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok, Thailand

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org